CLINICAL TRIAL: NCT07335055
Title: A Phase 2 Randomized, Double-blind, Placebo-Controlled, Multicenter Clinical Study to Evaluate the Efficacy and Safety of HSK47388 in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study for HSK47388 in Participants With Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK47388-202
Record Dates: First submitted 2026-01-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK47388-Dose level 1 (Experimental)
  Interventions: Drug: HSK47388
- HSK47388-Dose level 2 (Experimental)
  Interventions: Drug: HSK47388
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK47388 — Participants will be randomized to receive HSK47388, orally starting at Week 0 . At Week-12, all participants will be evaluated for clinical response and responders will enter the maintenance study.
  Arms: HSK47388-Dose level 1; HSK47388-Dose level 2
Drug: Placebo — Participants will be randomized to receive Placebo, orally starting at Week 0 . At Week-12, all participants will be evaluated for clinical response and responders will enter the maintenance study.
  Arms: Placebo

SUMMARY:
The purpose of this protocol is to evaluate the efficacy and safety of HSK47388 as therapy in participants with moderately to severely active ulcerative colitis .

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained
2. Male or female, ≥18 years old and ≤75 years old
3. Willing and able to comply with study-specific procedures and the requirements of study protocol.
4. Diagnosis of ulcerative colitis (UC)
5. Baseline modified Mayo score of 5 to 9 and the endoscopy subscore 2 to 3
6. Demonstrated an inadequate response, loss of response, or failure to tolerate previous conventional therapy or advanced therapy.

Exclusion Criteria:

1. Subjects have used treatments within the time frame specified in protocol prior to the baseline visit
2. Diagnosis of indeterminate colitis, ischemic colitis, Crohn's colitis or clinical findings suggestive of Crohn's disease
3. Participants with current or prior diagnosis of fulminant colitis and/or toxic megacolon
4. Presence of a stoma
5. Presence or history of a fistula
6. Intra-abdominal or other major surgery performed within 12 weeks before baseline
7. History of extensive colonic resection
8. Subjects have laboratory values meeting the criteria in protocol
9. Concurrent conditions and history of other diseases as described in protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with clinical response | Week 12

SECONDARY OUTCOMES:
The proportion of patients with clinical remission | Week 12
The proportion of patients with symptomatic remission | Week 12
The proportion of patients with endoscopic remission | Week 12
Proportion of patients with Mayo endoscopic subscore 0 | Week 12
Percent change from baseline in Mayo score and modified Mayo score | Week 12
Percent change from baseline in partial Mayo score | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided